CLINICAL TRIAL: NCT05182190
Title: Effects of Black Bean Pasta Consumption on Biomarkers in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Donna Winham, Assistant Professor, Food Science and Human Nutrition, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-191BB
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Glucose, High Blood
Keywords: glucose; insulin; legumes
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 5 x 5 crossover study with 3 treatments and two controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control - White bread (Active Comparator): Commercial white bread in a 50 gram available carbohydrate dose
  Interventions: Dietary Supplement: White bread
- Control - whole black beans (Active Comparator): Whole boiled black beans (Zenith) in a 50 gram available carbohydrate dose
  Interventions: Dietary Supplement: Black beans whole boiled
- Knife Mill pasta (Experimental): Heat treated black bean flour made with standard Knife Mill techniques
  Interventions: Dietary Supplement: Knife Mill pasta
- Combined pasta (Experimental): Black bean flour with medium protein made with novel compression/decompression mill
  Interventions: Dietary Supplement: Combo Flour Pasta
- Cyclone pasta (Experimental): Black bean flour with lower protein made with novel compression/decompression mill
  Interventions: Dietary Supplement: Cyclone Flour Pasta

INTERVENTIONS:
Dietary Supplement: White bread — Toasted white bread
  Arms: Control - White bread
Dietary Supplement: Black beans whole boiled — Whole boiled black beans with spaghetti sauce
  Arms: Control - whole black beans
Dietary Supplement: Knife Mill pasta — Black bean pasta (KM) with spaghetti sauce
  Arms: Knife Mill pasta
Dietary Supplement: Combo Flour Pasta — Black bean pasta (Combo) with spaghetti sauce (medium protein flour)
  Arms: Combined pasta
Dietary Supplement: Cyclone Flour Pasta — Black bean pasta (Cyclone) with spaghetti sauce (low protein flour)
  Arms: Cyclone pasta

SUMMARY:
The study purpose is to determine the effect of eating three (3) different pasta flour formulations made from 100% black beans (Zenith) in a meal matrix (spaghetti sauce) on postprandial glycemic response in healthy adults.

DETAILED DESCRIPTION:
The 5 test treatments (white bread (negative control), whole black beans (positive control), and 3 different pasta formulations) will be administered randomly over five weeks. Meals will be combined with spaghetti sauce for a total available carbohydrate amount of 50g.

Venous blood samples will be collected for glucose and insulin analysis at time 0 (fasting) and at 30, 60, 90, 120, and 180 minutes post-treatment (timing of the post-treatment blood draws started at time 0 [post-treatment], which is when the participant starts consuming the treatment meal). Blood analysis was completed by a reputable biomarker diagnostics laboratory, Quest Diagnostics.

Anthropometric measures such as weight, height, waist circumference, and blood pressure were collected at screening and at the start of each test day. Thirteen hours before testing, participants consumed a standardized frozen meal to reduce the potential variation in glycemic responses on test day due to varying pre-evening dietary intakes. This control meal was selected by each participant before the start of the study. Each participant was provided the same frozen meal every time, since the subjects serve as their own controls. The day before test day, participants completed a 24 hour food recall, satiety, and gastrointestinal questionnaires. The morning of each test day participants completed the International Physical Activity Questionnaire (IPAQ), satiety, and gastrointestinal questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* normal blood glucose
* BMI between 20-29.9 kg/m2.
* Chronic health conditions, e.g., hypertension, gastrointestinal disease.

Exclusion Criteria:

* Weight changes of >10% of body weight within previous 6 months
* Pregnant or breastfeeding
* Allergy to peas, beans, lentils, tomatoes, gluten, or latex
* Unwillingness or inability to follow study protocol

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in baseline blood glucose over 3 hours (glycemic response) | Time 0 (fasting) then every 30 minutes for 3 hours
  Venous blood samples were collected via venous catheter. Whole blood samples were analyzed for glucose content and insulin at commercial laboratory.

SECONDARY OUTCOMES:
Change in satiety sensation | Time 0 (fasting) then every 30 minutes for 3 hours
  Satiety level measured using a visual analog scale (0-100) every 30 minutes postprandially. A higher score indicates greater satiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Food Science and Human Nutrition Department, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No